CLINICAL TRIAL: NCT02922907
Title: Anti-Inflammatory Effects of Arabinoxylan Rice Bran Supplementation in Participants With Treated, Suppressed HIV Infection and Inadequate Immune Reconstitution
Brief Title: Rice Bran Supplementation in Treated HIV Infection
Acronym: BRM4
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Michael Dube, Professor of Medicine, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HS-16-00428
Record Dates: First submitted 2016-09-28; First posted 2016-10-04 (Estimated); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Inflammation in HIV Infection
MeSH Terms: interventions — polysaccharide MGN3

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arabinoxylan Rice Bran (Experimental): BRM4 two 500mg capsules thrice daily p.o. for 12 weeks
  Interventions: Dietary Supplement: arabinoxylan rice bran
- Placebo (Placebo Comparator): Placebo for BRM4 two 500mg capsules thrice daily p.o. for 12 weeks
  Interventions: Dietary Supplement: Placebo for arabinoxylan rice bran

INTERVENTIONS:
Dietary Supplement: arabinoxylan rice bran — a proprietary product derived from rice bran treated with extracts from three mushrooms
  Other Names: Biobran, BRM4
  Arms: Arabinoxylan Rice Bran
Dietary Supplement: Placebo for arabinoxylan rice bran — inactive product
  Arms: Placebo

SUMMARY:
Double-blind placebo-controlled randomized trial of Arabinoxylan Rice Bran Supplementation for 12 weeks with BRM4 in HIV-infected participants with inadequate immune reconstitution.

DETAILED DESCRIPTION:
Rationale: HIV infected persons have greater levels of inflammation and immune activation compared to the general population and are at greater risk of developing coronary heart disease (CHD) and other inflammation-associated co-morbidities. Intervention with BRM4 (Arabinoxylan Rice Bran Supplementation) in this population with impaired immune reconstitution may improve inflammation by a variety of mechanisms.

Intervention: Arabinoxylan Rice Bran Supplementation with BRM4, is a nutritional supplement marketed in the US. It is composed of dietary fiber obtained from a denatured hemicellulose that is obtained by reacting rice bran hemicellulose with multiple carbohydrate hydrolyzing enzymes from Shiitake mushrooms.

Objectives: The primary objective is to evaluate if 12 weeks of supplementation with arabinoxylan rice bran can safely reduce markers of inflammation during ART-suppressed HIV infection and thus potentially reduce the potential to develop end-organ disease in this group of at-risk patients.

Study population: HIV-infected participants (≥18 years of age) who have been on stable ART for at least 24 weeks prior to study entry, and have impaired immune reconstitution defined as a CD4+ T-cell count 100-350 cells/mm3 prior to study entry, with plasma HIV-1 RNA <50 copies/mL. In order to assure 24 evaluable subjects, the investigators will enroll 28 subjects total (assuming 15% lost to follow-up rate).

Study methodology: Randomized, double blind, placebo controlled clinical trial

Description of study arms: At entry participants will be randomized to one of the following arms:

Arm 1: BRM4 two 500mg capsules thrice daily p.o. for 12 weeks

Arm 2: Placebo for Biobran two capsules thrice daily p.o. for 12 weeks

Study endpoints: Primary - changes in sCD14 levels after 12 weeks of intervention. Secondary - week 12 changes in other inflammatory markers, microbial translocation, T-cell counts, and metabolic variables.

Follow-up: Participants will not be followed after study completion, unless follow-up is necessary for an adverse event.

Statistics: A total sample of 24 evaluable subjects (12 per arm) is needed to detect a clinically relevant difference of 0.07 log10 in sCD14 levels between treatment vs. placebo arms with 90% power and a 0.05 two-sided type I error rate.

Plans for analysis: For the primary analysis, changes in sCD14 (and other biomarkers) from baseline to week 12 will be compared between the treatment arm and the placebo arm by a two-sided, two-sample t-test.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV-1 infection
* Currently on a combination antiretroviral regimen for ≥24 weeks prior to study entry with no interruption longer than 7 consecutive days during that period.
* Plasma HIV-1 RNA levels below 50 copies/mL for at least 24 weeks prior to study entry.
* CD4+ cell count 100-350 cells/mm3 obtained within 90 days prior to study entry.
* The following laboratory values obtained within 90 days prior to entry by any US laboratory that has a CLIA certification or its equivalent.

  * Absolute neutrophil count (ANC) ≥750/mm3
  * Hemoglobin ≥8.0 g/dL
  * Platelet count ≥50,000/mm3
  * Calculated creatinine clearance (CrCl) ≥50 mL/min as estimated by the Cockroft-Gault formula
  * Aspartate aminotransferase (AST) (SGOT) ≤5 x upper limit of normal (ULN).
  * alanine aminotransferase (ALT) (SGPT) ≤5 x ULN.
  * alkaline phosphatase ≤5 x ULN.
  * Total bilirubin ≤2.5 x ULN (if the participant is receiving atazanavir, a total bilirubin of ≤5 x ULN is acceptable)
* For females of reproductive potential (women who have not been post-menopausal for at least 24 consecutive months, i.e. who have had menses within 24 months prior to study entry), or women who have not undergone surgical sterilization (specifically hysterectomy or bilateral oophorectomy or tubal ligation), will require a negative serum or urine pregnancy test (latter with a sensitivity of 15-25 mIU/mL) within 2 days prior to entry.
* If participating in sexual activity that could lead to pregnancy, the female study volunteer must be willing to use a contraceptive while receiving protocol-specified medication
* Men and women age 18 years or greater.
* Ability and willingness of participant or legal guardian/representative to provide informed consent.
* Participants on statin therapy must be stable on the same dose for at least the prior 12 weeks with no anticipated change in statin or dose during the intervention

Exclusion Criteria:

* Change in the ART regimen within the 12 weeks prior to study entry, or anticipated/intended modification of ART during the study period.
* Two or more HIV-1 RNA determinations >200 copies/mL within the 48 week period prior to study entry.
* Use of any immunomodulator, HIV vaccine, investigational therapy, or anti-TNF therapies within 90 days prior to study entry.
* Active malignancy with expected need for systemic chemotherapy or radiation therapy during the study period.
* Pregnant or breastfeeding.
* Known allergy/sensitivity to rice, rice bran, mushrooms, or related food products.
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Acute or serious illness requiring systemic treatment and/or hospitalization within 90 days prior to entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-03-24 (Actual); Primary Completion 2018-12-03 (Actual); Study Completion 2019-12-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in soluble CD14 levels will be compared between the supplement or placebo | 12 weeks
  Marker of macrophage activation

SECONDARY OUTCOMES:
Changes in LPS levels | 12 weeks
  measure of gut microbial translocation
changes in hsCRP levels | 12 weeks
  inflammatory biomarker
changes in D-dimer levels | 12 weeks
  coagulation biomarker
changes in soluble CD163 levels | 12 weeks
  marker of macrophage activation

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Dubé, MD, Study Director — University of Souther California
Locations (1):
- Rand Schrader Health and Research Clinic, Los Angeles, California, United States